CLINICAL TRIAL: NCT04102124
Title: A Phase II Clinical Study of SHR3680 Combined With SHR3162 in the Treatment of Metastatic Castration-resistant Prostate Cancer Previously Treated With Abiraterone and Docetaxel
Brief Title: A Study of SHR3680 in Combination With SHR3162 in the Treatment of mCRPC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor's R&D strategy is adjusted.
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR3680-SHR3162-II-CRPC
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer
Keywords: Castration-resistant Prostate Cancer; SHR3680; SHR3162
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR3680+SHR3162 (Experimental): Participants will receive SHR3680 combined with SHR3162 orally
  Interventions: Drug: SHR3680; Drug: SHR3162
- SHR3680+SHR3162(Placebo) (Experimental): Participants will receive SHR3680 combined with SHR3162(Placebo) orally
  Interventions: Drug: SHR3680; Drug: SHR3162(Placebo)
- SHR3680(Placebo)+SHR3162(Placebo) (Placebo Comparator): Participants will receive SHR3680(Placebo) combined with SHR3162(Placebo) orally
  Interventions: Drug: SHR3680(Placebo); Drug: SHR3162(Placebo)

INTERVENTIONS:
Drug: SHR3680 — Tablet. Specifications of 80mg
  Arms: SHR3680+SHR3162; SHR3680+SHR3162(Placebo)
Drug: SHR3162 — Tablet. Specifications of 10mg、40mg、50mg and 100mg
  Arms: SHR3680+SHR3162
Drug: SHR3680(Placebo) — Tablet. Specifications of 80mg
  Arms: SHR3680(Placebo)+SHR3162(Placebo)
Drug: SHR3162(Placebo) — Tablet. Specifications of 10mg、40mg、50mg and 100mg
  Arms: SHR3680(Placebo)+SHR3162(Placebo); SHR3680+SHR3162(Placebo)

SUMMARY:
The aim of this trial is to evaluate SHR3680 combined with SHR3162 and SHR3680 single drug to improve Metastatic Castration Resistant Prostate Cancer Patients whether the patient's overall survival (OS) is superior to placebo.

DETAILED DESCRIPTION:
This is a multicenter, randomized , double-blind Phase II trial and the aim of this trial is to evaluate SHR3680 combined with SHR3162 and SHR3680 single drug to improve Metastatic Castration Resistant Prostate Cancer Patients Previously Treated With Abiraterone and Docetaxel whether the patient's overall survival (OS) is superior to placebo. The Stage I part is a dose-escalation and -expansion study. Approximately 18~24 patients in Stage I will receive fixed-dose of orally SHR3680 and only one of two dose levels of orally SHR3162. The Primary endpoints of the Stage I are incidence of adverse events(AE) and recommended phase 2 dose(RP2D). The Stage II part is a randomized , double-blind study. Approximately 90~120 patients in Stage II will receive SHR3162 combined with SHR3680, in which one fixed-dose levels of SHR3162 will be selected based on the result of the Stage I.The Primary endpoint of the Stage II is overall survival(OS).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed prostate cancer; does not suggest neuroendocrine or small cell characteristics
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1;
3. Radiographic evidence of metastasis;
4. Sustained therapy of luteinizing hormone-releasing hormone analogue(LHRHA)or received bilateral orchiectomy; patients who did not receive bilateral orchiectomy are willing to receive sustained therapy of LHRHA;
5. Evidence of prostate cancer progression under the sustained therapy of LHRHA or bilateral orchiectomy;
6. Adequate hepatic, renal, heart, and hematological functions;
7. Patients have given voluntary written informed consent before performance of any study-related procedure not part of normal medical care,with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
8. Patient has been treated with Abiraterone and treatment failed（Treatment failure is defined as the progression of disease during treatment）
9. Patient has been treated with Docetaxel and treatment failed or can not tolerate docetaxel chemotherapy or patients who are not suitable for docetaxel treatment at the time of screening.

Exclusion Criteria:

1. Have received any anti-tumor therapy in the past 4 weeks,including radiotherapy, chemotherapy, operation, targeted therapy, immuntherapy, and endocrinotherapy;
2. Planned to initiate any other anti-tumor therapies during the study;
3. Unable to swallow, chronic diarrhea and intestinal obstruction, or the presence of a variety of other factors that affect drug use and absorption;
4. Clinically significant cardiovascular diseases;
5. History of seizure or certain conditions that may predispose to seizure;
6. Severe concurrent disease and infection that, in the judgment of the investigator, would make the patient inappropriate for enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse Event(AE) | Approximately 70 months
  The type, frequency, severity, timing, seriousness, and relationship to study therapy
Overall Survival(OS) | Approximately 70 months
  Time from randomisation to death due to any cause

SECONDARY OUTCOMES:
Time to prostate specific antigen (PSA) progression | Approximately 70 months
  Time from randomisation to the first time of PSA progression according to the criterion of PCGW3
Radiographic Progression Free Survival(rPFS) | Approximately 70 months
  Time from randomisation to radiologically confirmed progressive disease or death due to any cause
Objective response rate (ORR) | Approximately 70 months
  The percentage of patients with measureable disease at baseline who achieved a complete or partial response in their soft tissue disease using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
Time to skeletal-related events | Approximately 70 months
  Time from randomisation to the first occurrence of a skeletal-related event. The skeletal-related event is defined as the occurrence of either pathological or clinical fracture, spinal cord compression, bone-related radiotherapy or surgery.
PSA response rate | Approximately 70 months
  After the continuous therapy from randomisation to the end of the 12 weeks, the percentage of patients whose levels of PSA decreased by more than 50% compared with baseline.
Area Under the Curve (AUC) | Approximately 12 months
  The single dose and multiple dose PK will be calculated as data permits including AUC
Maximum Observed Plasma Concentration (Cmax) | Approximately 12 months
  The single-dose and multiple dose PK will be calculated as data permits including Cmax
Minimum Observed Plasma Concentration (Cmin) | Approximately 12 months
  The single-dose and multiple dose PK will be calculated as data permits including Cmin

CONTACTS AND LOCATIONS:
Locations (1):
- Ye Dingwei, Shanghai, China

IPD SHARING:
Plan to Share IPD: No